CLINICAL TRIAL: NCT05686239
Title: An Adaptive, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of RL-007 in the Treatment of Cognitive Impairment Associated With Schizophrenia (CIAS)
Brief Title: A Study to Evaluate RL-007 in the Treatment of Cognitive Impairment Associated With Schizophrenia (CIAS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recognify Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C07-03-02
Record Dates: First submitted 2022-12-28; First posted 2023-01-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment Associated With Schizophrenia (CIAS); Cognitive Impairment; Schizophrenia
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RL-007 20 mg (Inidascamine) (Experimental): oral dosing three times per day (TID)
  Interventions: Drug: RL-007 (Inidascamine)
- RL-007 40 mg (Inidascamine) (Experimental): oral dosing three times per day (TID)
  Interventions: Drug: RL-007 (Inidascamine)
- Placebo (Placebo Comparator): oral dosing three times per day (TID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RL-007 (Inidascamine) — investigational study drug
  Arms: RL-007 20 mg (Inidascamine); RL-007 40 mg (Inidascamine)
Drug: Placebo — placebo capsules matching the appearance and size of the active drug
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate if the investigational drug, RL-007, can improve the cognitive performance of subjects with schizophrenia. The main questions the study aims to answer are:

1. Does RL-007 improve subjects performance in a set of cognitive tasks?
2. Which dose of RL-007 (20 mg or 40 mg) has a larger effect on cognitive performance?
3. How well do subjects tolerate RL-007?

In the study, subjects will perform the cognitive tasks at the beginning to get familiar with the tasks. Then, subjects will be given either RL-007 or a placebo for 6 weeks and then repeat the cognitive tasks. The researchers will compare the results at the end of the treatment period to the baseline to see if there have been any changes in performance.

Additionally, several safety measures will be collected throughout the study (blood pressure, physical exam, ECGs, etc) to evaluate if there are any side effects from taking RL-007.

DETAILED DESCRIPTION:
This is a randomized, 3-arm, placebo-controlled, double-blinded clinical trial to evaluate the efficacy, safety, and tolerability of RL-007 in subjects with stable schizophrenia. The treatment period is 6 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of schizophrenia, per Diagnostic and Statistical Manual (DSM) 5, with a duration of at least 6 months
* Positive and Negative Symptoms Severity Score (PANSS) of less than or equal to 80 (inclusive)
* Currently treated on a single atypical antipsychotic (other than clozapine) at a stable dose and clinically stable for at least 6 weeks before randomization
* Clinical Global Impression - Severity score < 5.
* Body mass index (BMI) <= 40.0 kg/m^2 at screening
* Participant has reliable housing that is not expected to change during the study period with no expected significant life events that could affect study outcomes throughout entire study period.
* Sufficient fluency in English to understand and complete study instructions and assessments

Key Exclusion Criteria:

* History of hospitalization for medical indication or psychiatric hospitalization within 3 months prior to screening.
* Participants who present a serious risk of suicide, as evidenced by a) "yes" on items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) and meeting these criteria within the past 6 months, or b) posing a significant suicide risk in the Investigator's judgement.
* Participants who present a risk of serious harm to others, as evidence by any history within the past 2 years and any expressed homicidal ideation (with or without plan).
* Current diagnosis of another major psychiatric disorder, intellectual disability, or any major neurological disease, brain injury, epilepsy, or severe brain trauma.
* Evidence or history of significant cognitive impairment, other than associated with schizophrenia, that in the judgement of the Investigator or Sponsor would confound interpretation of study data or prevent safe and satisfactory completion of the study protocol.
* Meets criteria for moderate to severe substance/drug abuse disorder (including alcohol) per DSM-5 within the last 6 months prior to informed consent or a positive alcohol breath test or urine test for drugs of abuse at either Screening or Randomization Visits (except for benzodiazepines taken according to prescription and as an ongoing, stable regimen).
* Participant has undergone electroconvulsive therapy within the past 12 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery (MCCB) neurocognitive composite | 6 weeks
  change from baseline in composite of nine cognitive tests

SECONDARY OUTCOMES:
Symbol Coding | 6 weeks
  change from baseline
The Speed of Processing domain of the MCCB | 6 weeks
  change from baseline
The Attention/Vigilance domain of the MCCB | 6 weeks
  change from baseline
The Working Memory domain of the MCCB | 6 weeks
  change from baseline
The Verbal Memory domain of the MCCB | 6 weeks
  change from baseline
The Visual Learning domain of the MCCB | 6 weeks
  change from baseline
The Reasoning and Problem-solving domain of the MCCB | 6 weeks
  change from baseline
Clinical Global Impression - Severity (CGI-S) | 6 weeks
  change from baseline

OTHER OUTCOMES:
Safety measures | 6 weeks
  Treatment Emergent Adverse Events
The Virtual Reality Functional Capacity Assessment Tool (VRFCAT) | 6 weeks
  change from baseline
The Social Cognition domain of the MCCB | 6 weeks
  change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gary Walker, PhD, Study Director — Recognify Life Sciences
Locations (36):
- United States (20):
  - Recognify Research Site, Culver City, California
  - Collaborative Neuroscience Research, Garden Grove, California
  - Recognify Research Site, Lafayette, California
  - Recognify Research Site, Oceanside, California
  - Recognify Research Site, Orange, California
  - Recognify Research Site, Torrance, California
  - Recognify Research Site, Hialeah, Florida
  - Recognify Research Site, Miami, Florida
  - Recognify Research Site, Miami Lakes, Florida
  - Recognify Research Site, Atlanta, Georgia
  - Recognify Research Site, Augusta, Georgia
  - Recognify Research Site, Gaithersburg, Maryland
  - Recognify Research Site, Berlin, New Jersey
  - Recognify Research Site, Brooklyn, New York
  - Recognify Research Site, Chapel Hill, North Carolina
  - Recognify Research Site, Cincinnati, Ohio
  - Recognify Research Site, Cleveland, Ohio
  - Recognify Research Site, Dallas, Texas
  - Recognify Research Site, Houston, Texas
  - Recognify Research Site, Everett, Washington
- Bulgaria (7):
  - Recognify Research Site, Burgas
  - Recognify Research Site, Kardzhali
  - Recognify Research Site, Pleven
  - Recognify Research Site, Plovdiv
  - Recognify Research Site, Sofia
  - Recognify Research Site (a), Varna
  - Recognify Research Site (b), Varna
- Czechia (3):
  - Recognify Research Site, Pilsen
  - Recognify Research Site (a), Prague
  - Recognify Research Site (b), Prague
- Poland (6):
  - Recognify Research Site, Gdansk
  - Recognify Research Site, Gorlice
  - Recognify Research Site, Kielce
  - Recognify Research Site, Lodz
  - Recognify Research Site, Lublin
  - Recognify Research Site, Poznan

IPD SHARING:
Plan to Share IPD: No